CLINICAL TRIAL: NCT03630276
Title: Evaluation of Neutrophil/Lymphocyte Ratio, Platelet /Lymphocyte Ratio and CRP as Markers of Severity of Pre-eclampsia
Brief Title: Evaluation of Neutrophil/Lymphocyte Ratio ,Platelet/Lymphocyte Ratio and CRP as Markers of Severity of Pre-eclampsia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Shaza Mohamed Elreweny, Shaza Mohamed Elreweny, Ain Shams University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: Shaza Elreweny
Record Dates: First submitted 2018-08-10; First posted 2018-08-14 (Actual); Last update posted 2018-08-14 (Actual); Status verified 2018-08

CONDITIONS: Pre-Eclampsia
MeSH Terms: conditions — Pre-Eclampsia | interventions — Platelet Count

STUDY DESIGN:
Who Masked: Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Neutrophil/lymphocyte ratio (Other)
  Interventions: Diagnostic Test: Neutrophil/lymphocyte ratio, Platelet /lymphocyte ratio and CRP
- Platelet/lymphocyte ratio (Other)
  Interventions: Diagnostic Test: Neutrophil/lymphocyte ratio, Platelet /lymphocyte ratio and CRP
- CRP (Other)
  Interventions: Diagnostic Test: Neutrophil/lymphocyte ratio, Platelet /lymphocyte ratio and CRP

INTERVENTIONS:
Diagnostic Test: Neutrophil/lymphocyte ratio, Platelet /lymphocyte ratio and CRP — Lab

SUMMARY:
Evaluation of neutrophil/lymphocyte ratio, Platelet /lymphocyte ratio and CRP as markers of severity of Pre-eclampsia

ELIGIBILITY:
Inclusion Criteria:

- PREECLAMPSIA from 25_45years

Exclusion Criteria:

* chronic diseases Primary hypertension

Ages: 25 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 111 (Estimated)
Dates: Start 2018-08-01 (Actual); Primary Completion 2018-08-10 (Actual); Study Completion 2018-08-10 (Estimated)

PRIMARY OUTCOMES:
PREECLAMPSIA | 6months

CONTACTS AND LOCATIONS:
Locations (1):
- Shaza, Alexandria, Alex, Egypt